CLINICAL TRIAL: NCT03807882
Title: Comparison of Maintenance ECT Versus Clozapine on Psychopathology and Cerebral Hemodynamics in Treatment-resistant Schizophrenia: A Randomized Controlled Trial
Brief Title: Comparison of Maintenance ECT Versus Clozapine in Treatment-resistant Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, BISWA RANJAN MISHRA, ADDITIONAL PROFESSOR, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T/IM-F/18-19/08
Record Dates: First submitted 2018-11-28; First posted 2019-01-17 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Treatment Resistant Schizophrenia
Keywords: M-ECT; Clozapine; Psychopathology; Cerebral perfusion
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant | interventions — Clozapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Bilateral Maintenance ECT (B/L M-ECT)
  Interventions: Other: Bilateral M-ECT
- Control group (Active Comparator): Clozapine monotherapy. Clozapine will be given in accordance with Maudsley guideline: 12.5 mg on the first day, followed by 12.5mg twice daily on the second day, followed by 25mg twice daily for next two days and then increment of 25mg every two days till the target dose of 250-400 mg per day in two divided doses as per tolerability of the patients
  Interventions: Drug: Clozapine

INTERVENTIONS:
Other: Bilateral M-ECT — Following acute treatment with bilateral ECT of 6 sessions over a period of two weeks, Bilateral M-ECT will be administered at a frequency of 1 session/week for one month, then 1 session / 2 weeks for 2 months and then 1 session/month for next 3 months.
  Arms: Test group
Drug: Clozapine — Clozapine will be given in accordance with Maudsley guideline: 12.5 mg on the first day, followed by 12.5mg twice daily on the second day, followed by 25mg twice daily for next two days and then increment of 25mg every two days till the target dose of 250-400 mg per day in two divided doses as per tolerability of the patients
  Arms: Control group

SUMMARY:
The proposed study will be conducted to compare the efficacy of maintenance ECT (M-ECT) vs Clozapine in treatment resistant schizophrenia (TRS) in terms of change in psychopathology measures and cerebral hemodynamics.

DETAILED DESCRIPTION:
The proposed study is a prospective, randomized clinical trial in patients suffering from treatment-resistant schizophrenia (TRS) and will be conducted in the Department of Psychiatry, AIIMS, Bhubaneswar, over a period of 16 months. Sixty patients with TRS (TRRIP consensus criteria, 2017), fulfilling the inclusion and exclusion criteria will be recruited for the study. Written informed consent will be taken after explaining the objectives and procedure of the study in detail. The detailed history, relevant social-demographic and clinical data will be collected in a structured case record form (CRF). At baseline, PANSS will be administered to determine the severity of positive symptoms, negative symptoms, and general psychopathology, Global assessment of functioning (GAF), and CGI to determine the baseline severity of the illness and improvement with treatment and MoCA to assess change in cognitive impairment. Before starting the treatment, brain SPECT-CT will be done to measure baseline regional brain blood perfusion. The study cohort will be randomized into two treatment groups by computer-generated random numbers, each group comprising 30 patients. One group will receive maintenance ECT (M-ECT) following acute treatment of bilateral ECT of six sessions along with ongoing antipsychotic and the other group will be treated with Clozapine monotherapy. PANSS, GAF, CGI, MoCA will be re-administered at 6 weeks, 3 months, and 6 months follow-up visits to compare the changes within each group and between the groups. Post-treatment SPECT-CT of the brain will be done at the end of 6 months to document changes in the regional cerebral blood perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed with treatment-resistant schizophrenia (TRS) (TRRIP consensus criteria).
* Patients aged 18-60 years of either sex.
* Patients giving voluntary written consent for participation in the study

Exclusion Criteria:

* Patient already on Clozapine or ECT.
* History of psychoactive substance abuse or dependence.
* Co-morbid psychiatric, major medical, or neurological disorders.
* History of organicity or significant head injury.
* Pacemaker or metal in any part of the body excluding the mouth.
* Pregnant and breastfeeding females.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in severity of psychopathology | 24 weeks
  Severity will be assessed by Positive and Negative Symptom Scale (PANSS) PANSS Score ranges from 30- 210. A higher score represents more severe psychopathology

SECONDARY OUTCOMES:
Change in illness severity, and global improvement with treatment | 24 weeks
  Assessed by change in Clinical Global Impression Schizophrenia (CGI-SCH) scores.
Change in global functionality | 24 weeks
  Assessed by change in Global assessment of functioning (GAF) scores.
Change in Cognitive impairment | 24 weeks
  Assessed by change in Montreal Cognitive Assessment (MoCA) scores.
Number of patients receiving rescue medications. | 24 weeks
  Patients with "treatment relapse" or "treatment non-response" will receive rescue medications.
Change in regional cerebral blood flow | 24 weeks
  Change in regional cerebral blood flow will be measured by SPECT-CT Brain

CONTACTS AND LOCATIONS:
Overall Officials: RITUPARNA MAITI, M.D, Study Chair — AIIMS Bhubaneswar
Locations (1):
- Dept of Psychiatry, Aiims, Bhubaneswar, Bhubaneswar, Odisha, India

REFERENCES:
- [Result] Kane JM. Management strategies for the treatment of schizophrenia. J Clin Psychiatry. 1999;60 Suppl 12:13-7. PMID 10372604
- [Result] Lieberman JA. Maximizing clozapine therapy: managing side effects. J Clin Psychiatry. 1998;59 Suppl 3:38-43. PMID 9541337
- [Result] Kim HS, Kim SH, Lee NY, Youn T, Lee JH, Chung S, Kim YS, Chung IW. Effectiveness of Electroconvulsive Therapy Augmentation on Clozapine-Resistant Schizophrenia. Psychiatry Investig. 2017 Jan;14(1):58-62. doi: 10.4306/pi.2017.14.1.58. Epub 2016 Dec 29. PMID 28096876
- [Result] Rey JM, Walter G. Half a century of ECT use in young people. Am J Psychiatry. 1997 May;154(5):595-602. doi: 10.1176/ajp.154.5.595. PMID 9137112
- [Result] Chanpattana W, Andrade C. ECT for treatment-resistant schizophrenia: a response from the far East to the UK. NICE report. J ECT. 2006 Mar;22(1):4-12. doi: 10.1097/00124509-200603000-00002. PMID 16633199
- [Result] Chanpattana W, Chakrabhand ML, Sackeim HA, Kitaroonchai W, Kongsakon R, Techakasem P, Buppanharun W, Tuntirungsee Y, Kirdcharoen N. Continuation ECT in treatment-resistant schizophrenia: a controlled study. J ECT. 1999 Sep;15(3):178-92. PMID 10492856
- [Result] Shimizu E, Imai M, Fujisaki M, Shinoda N, Handa S, Watanabe H, Nakazato M, Hashimoto K, Iyo M. Maintenance electroconvulsive therapy (ECT) for treatment-resistant disorganized schizophrenia. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Mar 30;31(2):571-3. doi: 10.1016/j.pnpbp.2006.11.014. Epub 2006 Dec 20. PMID 17187911
- [Result] Grover S, Hazari N, Kate N. Combined use of clozapine and ECT: a review. Acta Neuropsychiatr. 2015 Jun;27(3):131-42. doi: 10.1017/neu.2015.8. Epub 2015 Feb 20. PMID 25697225
- [Result] Petrides G, Malur C, Braga RJ, Bailine SH, Schooler NR, Malhotra AK, Kane JM, Sanghani S, Goldberg TE, John M, Mendelowitz A. Electroconvulsive therapy augmentation in clozapine-resistant schizophrenia: a prospective, randomized study. Am J Psychiatry. 2015 Jan;172(1):52-8. doi: 10.1176/appi.ajp.2014.13060787. Epub 2014 Oct 31. PMID 25157964
- [Result] Lally J, Tully J, Robertson D, Stubbs B, Gaughran F, MacCabe JH. Augmentation of clozapine with electroconvulsive therapy in treatment resistant schizophrenia: A systematic review and meta-analysis. Schizophr Res. 2016 Mar;171(1-3):215-24. doi: 10.1016/j.schres.2016.01.024. Epub 2016 Jan 27. PMID 26827129
- [Result] Siskind DJ, Lee M, Ravindran A, Zhang Q, Ma E, Motamarri B, Kisely S. Augmentation strategies for clozapine refractory schizophrenia: A systematic review and meta-analysis. Aust N Z J Psychiatry. 2018 Aug;52(8):751-767. doi: 10.1177/0004867418772351. Epub 2018 May 6. PMID 29732913
- [Result] Santra A, Kumar R. Brain perfusion single photon emission computed tomography in major psychiatric disorders: From basics to clinical practice. Indian J Nucl Med. 2014 Oct;29(4):210-21. doi: 10.4103/0972-3919.142622. PMID 25400359
- [Result] Ertugrul A, Volkan-Salanci B, Basar K, Karli Oguz K, Demir B, Ergun EL, Senturk S, Erbas B, Cila A, Ulug B. The effect of clozapine on regional cerebral blood flow and brain metabolite ratios in schizophrenia: relationship with treatment response. Psychiatry Res. 2009 Nov 30;174(2):121-9. doi: 10.1016/j.pscychresns.2009.04.007. Epub 2009 Oct 17. PMID 19837567
- [Result] Novak B, Milcinski M, Grmek M, Kocmur M. Early effects of treatment on regional cerebral blood flow in first episode schizophrenia patients evaluated with 99Tc-ECD-SPECT. Neuro Endocrinol Lett. 2005 Dec;26(6):685-9. PMID 16380684
- [Result] Sharafi M. Comparison of Classical and Clozapine Treatment on Schizophrenia Using Positive and Negative Syndrome Scale of Schizophrenia (PANSS) and SPECT Imaging. Int J Med Sci. 2005;2(2):79-86. doi: 10.7150/ijms.2.79. Epub 2005 May 10. PMID 15968344
- [Result] Howes OD, McCutcheon R, Agid O, de Bartolomeis A, van Beveren NJ, Birnbaum ML, Bloomfield MA, Bressan RA, Buchanan RW, Carpenter WT, Castle DJ, Citrome L, Daskalakis ZJ, Davidson M, Drake RJ, Dursun S, Ebdrup BH, Elkis H, Falkai P, Fleischacker WW, Gadelha A, Gaughran F, Glenthoj BY, Graff-Guerrero A, Hallak JE, Honer WG, Kennedy J, Kinon BJ, Lawrie SM, Lee J, Leweke FM, MacCabe JH, McNabb CB, Meltzer H, Moller HJ, Nakajima S, Pantelis C, Reis Marques T, Remington G, Rossell SL, Russell BR, Siu CO, Suzuki T, Sommer IE, Taylor D, Thomas N, Ucok A, Umbricht D, Walters JT, Kane J, Correll CU. Treatment-Resistant Schizophrenia: Treatment Response and Resistance in Psychosis (TRRIP) Working Group Consensus Guidelines on Diagnosis and Terminology. Am J Psychiatry. 2017 Mar 1;174(3):216-229. doi: 10.1176/appi.ajp.2016.16050503. Epub 2016 Dec 6. PMID 27919182
- [Derived] Mishra BR, Agrawal K, Biswas T, Mohapatra D, Nath S, Maiti R. Comparison of Acute Followed by Maintenance ECT vs Clozapine on Psychopathology and Regional Cerebral Blood Flow in Treatment-Resistant Schizophrenia: A Randomized Controlled Trial. Schizophr Bull. 2022 Jun 21;48(4):814-825. doi: 10.1093/schbul/sbac027. PMID 35556138